CLINICAL TRIAL: NCT04282785
Title: Point-of-care Monitoring of Antibiotic Concentration in Blood With UV-VIS Absorption Spectroscopy
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: ABABS001
Record Dates: First submitted 2019-04-18; First posted 2020-02-25 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Infection, Bacterial
Keywords: meropenem; cefotaxime; piperacillin/tazobactam; Drug Monitoring; Antibiotics
MeSH Terms: conditions — Sepsis; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort of patients with severe infections: Patients with severe infections admitted to the Uppsala University Hospital and gets treated with either Piperacillin-Tazobactam, Meropenem or Cefotaxim
  Interventions: Diagnostic Test: Concentration monitoring of antibiotics in plasma

INTERVENTIONS:
Diagnostic Test: Concentration monitoring of antibiotics in plasma — Plasma antibiotic concentration will be measured using a bedside method with UV-VIS spectroscopy. These measurements will be validated with golden standard that is HPLC-MS.

SUMMARY:
This prospective clinical study will investigate if antibiotic concentrations in patients with severe infections can be monitored by the UV-VIS spectroscopy.

DETAILED DESCRIPTION:
Early and correct antibiotic treatment has a fundamental effect on survival in severe infections, and to prevent resistance development. However, it is unclear if this is achieved in severely ill patients with severe infections. Underdosing of antibiotics leads to lack of effect against bacteria and selection of multi-resistant strains. Overdosing of antibiotics increases the risk of toxicity and poses a threat to the environment. Currently there is no method for rapid or bedside determination of antibiotic concentration in routine health care.

Pharmacolog AB, an Uppsala Med-tech company, has developed a technology and a product DrugLog® based on absorption spectroscopy in ultraviolet - visible (UV-VIS) frequencies that can measure the concentration of antibiotics.

The goal of this project is to investigate if antibiotic concentrations in patients could be monitored by the UV-VIS spectroscopy.

In a prospective observational study, blood samples from 100 patients with severe infections treated with cefotaxime, piperacillin/tazobactam or meropenem will be measured by UV-VIS spectroscopy as well as with the golden standard, High-performance liquid chromatography-mass spectrometry (HPLC-MS) at Klinisk farmakologi, Huddinge hospital, Stockholm.

After informed consent, samples will be taken prior to antibiotic treatment and three times thereafter. Demographic and clinical data will be registered.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Suspected infection where treatment with cefotaxime, piperacillin/tazobactam or meropenem is prescribed

Exclusion Criteria:

* Pregnancy
* Intermittent haemodialysis
* Patient with limited treatment decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients with suspected infection that is prescribed with antibiotics (cefotaxime, piperacillin/tazobactam or meropenem) that is hospitalized and admitted to the infection ward, Intermediate ward or ICU.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Agreement in antibiotic concentration in blood with UV-VIS technique vs. HPLC-MS expressed bias (limits of agreements) in a Bland Altman plot. | 0-48 hours of antibiotic treatment.
  The antibiotic concentration will be calculated from the change in from transmittance measured with UV-VIS spectroscopy technique and compared with change antibiotic concentration measured with HPLC-MS using linear regression and Bland-Altman plots. The endpoint will be presented as bias (limits of agreement).

SECONDARY OUTCOMES:
Agreement in antibiotic concentration change in blood after antibiotic administration with UV-VIS technique vs HPLC-MS | Blood samples will be taken just before the first dose of antibiotic, two hours after the first dose of antibiotic, just before the second dose and two hours after the second dose.
  The antibiotic concentration will be calculated from the change in from transmittance measured with UV-VIS spectroscopy technique and compared with change antibiotic concentration measured with HPLC-MS using linear regression and Bland-Altman plots. The endpoint will be presented as bias (limits of agreement).

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Lipcsey, Principal Investigator — Department of surgical science, Uppsala University hospital
Locations (1):
- Uppsala university hospital, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Background] Bagshaw SM, Lapinsky S, Dial S, Arabi Y, Dodek P, Wood G, Ellis P, Guzman J, Marshall J, Parrillo JE, Skrobik Y, Kumar A; Cooperative Antimicrobial Therapy of Septic Shock (CATSS) Database Research Group. Acute kidney injury in septic shock: clinical outcomes and impact of duration of hypotension prior to initiation of antimicrobial therapy. Intensive Care Med. 2009 May;35(5):871-81. doi: 10.1007/s00134-008-1367-2. Epub 2008 Dec 9. PMID 19066848
- [Background] Brink AJ, Richards GA, Schillack V, Kiem S, Schentag J. Pharmacokinetics of once-daily dosing of ertapenem in critically ill patients with severe sepsis. Int J Antimicrob Agents. 2009 May;33(5):432-6. doi: 10.1016/j.ijantimicag.2008.10.005. Epub 2008 Dec 16. PMID 19091521
- [Background] Fuchs M, Sanyal AJ. Sepsis and cholestasis. Clin Liver Dis. 2008 Feb;12(1):151-72, ix. doi: 10.1016/j.cld.2007.11.002. PMID 18242502
- [Background] Garot D, Respaud R, Lanotte P, Simon N, Mercier E, Ehrmann S, Perrotin D, Dequin PF, Le Guellec C. Population pharmacokinetics of ceftriaxone in critically ill septic patients: a reappraisal. Br J Clin Pharmacol. 2011 Nov;72(5):758-67. doi: 10.1111/j.1365-2125.2011.04005.x. PMID 21545483
- [Background] Green L, Dick JD, Goldberger SP, Angelopulos CM. Prolonged elimination of piperacillin in a patient with renal and liver failure. Drug Intell Clin Pharm. 1985 Jun;19(6):427-9. doi: 10.1177/106002808501900604. PMID 4006736
- [Background] SAFE Study Investigators; Finfer S, McEvoy S, Bellomo R, McArthur C, Myburgh J, Norton R. Impact of albumin compared to saline on organ function and mortality of patients with severe sepsis. Intensive Care Med. 2011 Jan;37(1):86-96. doi: 10.1007/s00134-010-2039-6. Epub 2010 Oct 6. PMID 20924555
- [Background] Jager NG, van Hest RM, Lipman J, Taccone FS, Roberts JA. Therapeutic drug monitoring of anti-infective agents in critically ill patients. Expert Rev Clin Pharmacol. 2016 Jul;9(7):961-79. doi: 10.1586/17512433.2016.1172209. Epub 2016 Apr 15. PMID 27018631
- [Background] Kieft H, Hoepelman AI, Knupp CA, van Dijk A, Branger JM, Struyvenberg A, Verhoef J. Pharmacokinetics of cefepime in patients with the sepsis syndrome. J Antimicrob Chemother. 1993 Nov;32 Suppl B:117-22. doi: 10.1093/jac/32.suppl_b.117. PMID 8150754
- [Background] Kumar A, Roberts D, Wood KE, Light B, Parrillo JE, Sharma S, Suppes R, Feinstein D, Zanotti S, Taiberg L, Gurka D, Kumar A, Cheang M. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006 Jun;34(6):1589-96. doi: 10.1097/01.CCM.0000217961.75225.E9. PMID 16625125
- [Background] Lau AH, Kronfol NO, John E. Increased vancomycin elimination with continuous hemofiltration. ASAIO Trans. 1987 Jul-Sep;33(3):772-4. No abstract available. PMID 3676016
- [Background] Liu KD, Thompson BT, Ancukiewicz M, Steingrub JS, Douglas IS, Matthay MA, Wright P, Peterson MW, Rock P, Hyzy RC, Anzueto A, Truwit JD; National Institutes of Health National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome Network. Acute kidney injury in patients with acute lung injury: impact of fluid accumulation on classification of acute kidney injury and associated outcomes. Crit Care Med. 2011 Dec;39(12):2665-71. doi: 10.1097/CCM.0b013e318228234b. PMID 21785346
- [Background] Macnab MS, Macrae DJ, Guy E, Grant IS, Feely J. Profound reduction in morphine clearance and liver blood flow in shock. Intensive Care Med. 1986;12(5):366-9. doi: 10.1007/BF00292927. PMID 3771915
- [Background] Roberts DM, Roberts JA, Roberts MS, Liu X, Nair P, Cole L, Lipman J, Bellomo R; RENAL Replacement Therapy Study Investigators. Variability of antibiotic concentrations in critically ill patients receiving continuous renal replacement therapy: a multicentre pharmacokinetic study. Crit Care Med. 2012 May;40(5):1523-8. doi: 10.1097/CCM.0b013e318241e553. PMID 22511133
- [Background] Roberts JA, Paul SK, Akova M, Bassetti M, De Waele JJ, Dimopoulos G, Kaukonen KM, Koulenti D, Martin C, Montravers P, Rello J, Rhodes A, Starr T, Wallis SC, Lipman J; DALI Study. DALI: defining antibiotic levels in intensive care unit patients: are current beta-lactam antibiotic doses sufficient for critically ill patients? Clin Infect Dis. 2014 Apr;58(8):1072-83. doi: 10.1093/cid/ciu027. Epub 2014 Jan 14. PMID 24429437
- [Background] Salam FA, Shoaib MH, Yousuf RI, Sultan F, Khan MA, Manzoor S. Simultaneous quantitation of Ofloxacin, Fexofenadine HCl and Diclofenac Potassium in affixed dose combinative formulation by HPLC-UV method. Pak J Pharm Sci. 2015 Nov;28(6):1979-84. PMID 26639475
- [Background] Sime FB, Udy AA, Roberts JA. Augmented renal clearance in critically ill patients: etiology, definition and implications for beta-lactam dose optimization. Curr Opin Pharmacol. 2015 Oct;24:1-6. doi: 10.1016/j.coph.2015.06.002. Epub 2015 Jun 25. PMID 26119486
- [Background] Wen X, Peng Z, Kellum JA. Pathogenesis of acute kidney injury: effects of remote tissue damage on the kidney. Contrib Nephrol. 2011;174:129-137. doi: 10.1159/000329382. Epub 2011 Sep 9. PMID 21921617
- [Background] White LE, Hassoun HT, Bihorac A, Moore LJ, Sailors RM, McKinley BA, Valdivia A, Moore FA. Acute kidney injury is surprisingly common and a powerful predictor of mortality in surgical sepsis. J Trauma Acute Care Surg. 2013 Sep;75(3):432-8. doi: 10.1097/TA.0b013e31829de6cd. PMID 24089113
- [Background] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Background] Wolff F, Deprez G, Seyler L, Taccone F, Hites M, Gulbis B, Vincent JL, Jacobs F, Cotton F. Rapid quantification of six beta-lactams to optimize dosage regimens in severely septic patients. Talanta. 2013 Jan 15;103:153-60. doi: 10.1016/j.talanta.2012.10.024. Epub 2012 Oct 18. PMID 23200371